CLINICAL TRIAL: NCT00798213
Title: A Phase 2 Study of SCH 727965 in Subjects With Relapsed and Refractory Acute Myelogenous Leukemia and Acute Lymphoblastic Leukemia
Brief Title: SCH 727965 in Patients With Acute Myelogenous Leukemia and Acute Lymphoblastic Leukemia (P04717AM2)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04717
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Leukemia, Myeloid, Acute; Lymphoblastic Leukemia, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — dinaciclib; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Participants with AML randomized to SCH 727965 (Experimental)
  Interventions: Drug: SCH 727965
- Participants with AML randomized to gemtuzumab ozogamicin (Active Comparator)
  Interventions: Drug: Gemtuzumab ozogamicin
- AML treated w/ SCH 727965 after prog. on gemtuzumab ozogamicin (Experimental)
  Interventions: Drug: SCH 727965
- Participants with ALL treated with SCH 727965 (Experimental)
  Interventions: Drug: SCH 727965

INTERVENTIONS:
Drug: SCH 727965 — SCH 727965 50 mg/m2 IV on Day 1 of each 21 day cycle until disease progression.
  Arms: AML treated w/ SCH 727965 after prog. on gemtuzumab ozogamicin; Participants with ALL treated with SCH 727965; Participants with AML randomized to SCH 727965
Drug: Gemtuzumab ozogamicin — Gemtuzumab ozogamicin 9 mg/m2 IV on Day 1 and Day 15.
  Other Names: Mylotarg
  Arms: Participants with AML randomized to gemtuzumab ozogamicin

SUMMARY:
Participants with acute myelogenous leukemia (AML) will be randomized to SCH 727965 or gemtuzumab ozogamicin. All participants with acute lymphoblastic leukemia (ALL) will receive SCH 727965. Part 1 of the study will determine the activity of SCH 727965 treatment in participants with AML and participants with ALL. Part 2 of the study will determine the activity of SCH 727965 treatment in participants with AML who experienced disease progression after standard treatment with gemtuzumab ozogamicin during Part 1.

ELIGIBILITY:
Inclusion Criteria:

* For participants with AML:

  * Age >=60 years, either sex, any race.
  * Diagnosis of CD33-positive AML by World Health Organization criteria.
  * Must be in first or second relapse, or have primary refractory or refractory disease at first salvage, and not be considered a candidate for transplant.
  * Acute promyelocytic leukemia who has relapsed following treatment with both all trans retinoic acid (tretinoin) and arsenic trioxide-based therapy is eligible.
* For participants with ALL:

  * Age >=18 years, either sex, any race.
  * Diagnosis of ALL by World Health Organization criteria.
  * Must be in first or second relapse, or have primary refractory or refractory disease at first salvage, and not be considered a candidate for potentially curative therapy.
  * Eastern Cooperative Oncology group performance status of 0 or 1.
  * Adequate hematologic, renal, and hepatic organ function and laboratory parameters.
  * Receiving treatment with hydroxyurea or leukapheresis to reduce elevated white blood cell count to <=30 x 10^9 is eligible, provided hydroxyurea and leukapheresis are discontinued at least 24 hours before initiation of study drug.

Exclusion Criteria:

* Known central nervous system leukemia.
* Previous hematopoietic stem cell transplantation.
* Previous treatment with SCH 727965 or other cyclin-dependent kinase inhibitors.
* For AML, previous treatment with gemtuzumab ozogamicin.
* Known HIV infection.
* Known active hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate of initial treatment with SCH 727965 in subjects with AML or ALL. | Time to identified response or disease progression on SCH 727965 in Part 1 (approx. 5 months).
Overall response rate in participants with AML treated with SCH 727965 after disease progression on comparator. | Time to identified response or disease progression on SCH 727965 in Part 2 (approx. 5 months).

SECONDARY OUTCOMES:
Time to disease progression for initial treatment with SCH 727965 in subjects with AML or ALL. | Time to identified disease progression on SCH 727965 in Part 1 (approx. 5 months).
Overall response rate and time to progression of treatment with gemtuzumab ozogamicin in subjects with AML. | Time to identified response or disease progression on gemtuzumab ozogamicin (approx. 5 months).
Time to disease progression for treatment with gemtuzumab ozogamicin in participants with AML. | Time to identified disease progression on gemtuzumab ozogamicin (approx. 5 months).
Time to disease progression in participants with AML treated with SCH 727965 after disease progression on gemtuzumab ozogamicin | Time to identified disease progression on SCH 727965 in Part 2 (approx. 5 months).

REFERENCES:
- [Result] Gojo I, Sadowska M, Walker A, Feldman EJ, Iyer SP, Baer MR, Sausville EA, Lapidus RG, Zhang D, Zhu Y, Jou YM, Poon J, Small K, Bannerji R. Clinical and laboratory studies of the novel cyclin-dependent kinase inhibitor dinaciclib (SCH 727965) in acute leukemias. Cancer Chemother Pharmacol. 2013 Oct;72(4):897-908. doi: 10.1007/s00280-013-2249-z. Epub 2013 Aug 15. PMID 23949430